CLINICAL TRIAL: NCT01443572
Title: The Comparison of Desflurane and Sevoflurane on Postoperative Recovery and Hepatic Function of Biliary Atresia Patients During Kasai Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2011-0436
Record Dates: First submitted 2011-09-16; First posted 2011-09-29 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Kasai Operation; Biliary Atresia
Keywords: Kasai operation under general anesthesia
MeSH Terms: conditions — Biliary Atresia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- desflurane group (Experimental)
  Interventions: Drug: desflurane anesthetics
- sevoflurane group (Active Comparator)
  Interventions: Drug: sevoflurane anesthetics

INTERVENTIONS:
Drug: desflurane anesthetics — 40 patients are randomly allocated into two groups : desflurane group (n=20) and sevoflurane group (n=20). And anesthesia is maintained with desflurane (desflurane group) or sevoflurane (sevoflurane group).
  Arms: desflurane group
Drug: sevoflurane anesthetics — 40 patients are randomly allocated into two groups : desflurane group (n=20) and sevoflurane group (n=20). And anesthesia is maintained with desflurane (desflurane group) or sevoflurane (sevoflurane group).
  Arms: sevoflurane group

SUMMARY:
Biliary atresia (BA) is a perinatal disease of unclear etiology, characterized by inflammation and obliteration of intrahepatic and extrahepatic bile ducts, leading to cholestasis and cirrhosis. Kasai operation remains as the first line operative treatment in BA. In the previous studies, inhalation anesthetics might induce liver damage. The choice of inhalation anesthetic that minimally affects hepatic function is important. Therefore, the purpose of this study is to compare the postoperative recovery and hepatic function between desflurane and sevoflurane, two most frequently used inhalational anesthetics in patients undergoing Kasai operation.

ELIGIBILITY:
Inclusion Criteria:

* patients with biliary atresia undergoing Kasai operation

Exclusion Criteria:

* patients with congenital anomalies at major organs

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in postoperative recovery | after operation, and on the 1st, 2nd, 3rd, 5th, 7th and 15th postoperative days.
  Complete blood count(CBC), prothrombin time(PT), activated partial thromboplastin time(APTT), aspartate aminotransferase(AST), alanine aminotransferase(ALT), alkaline phosphatase(ALP), albumin, total bilirubin, direct bilirubin, gamma-GTP, BUN, creatinine(Cr), electrolyte
Change in hepatic function | after operation, and on the 1st, 2nd, 3rd, 5th, 7th and 15th postoperative days
  Complete blood count(CBC), prothrombin time(PT), activated partial thromboplastin time(APTT), aspartate aminotransferase(AST), alanine aminotransferase(ALT), alkaline phosphatase(ALP), albumin, total bilirubin, direct bilirubin, gamma-GTP, BUN, creatinine(Cr), electrolyte

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea